CLINICAL TRIAL: NCT06366867
Title: An Open Platform of Serious Games for Cognitive Intervention
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Technical issues
Sponsor: University of Alberta (Other)
Collaborators: Alberta Health services (Other); CapitalCare (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Device Feasibility
Other Study IDs: Pro00097579
Record Dates: First submitted 2024-04-04; First posted 2024-04-16 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Mild Cognitive Impairment; Dementia; Alzheimer Disease; Aging
Keywords: Serious computer game; computer games; VibrantMinds
MeSH Terms: conditions — Cognitive Dysfunction; Dementia; Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: The experimental group will receive VibrantMinds, which consists of sessions with serious computer games in addition to the standard care, whilst the control group will receive the standard of care used at the healthcare facilities.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Random allocation, 1:1 ratio by a computer-based randomizer
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VibrantMinds + Standard Care (Experimental): Older adults at long-term care facilities receive the VibrantMinds games in addition to routine standard care administered by the facility and staff.
  Interventions: Device: VibrantMinds
- Standard Care (No Intervention): Older adults at long-term care facilities receive routine standard care administered by the facility and staff.

INTERVENTIONS:
Device: VibrantMinds — VibrantMindVibrantMinds offers five tablet games targeting cognitive stimulation in older adults: Whack-A-Mole, Word Search, Bejeweled, Mahjong Solitaire, Memory Game, and Glenrose Grocery Game (GGG). These games vary from nostalgic (e.g., Mahjong Solitaire) to leisure-oriented (e.g., Bejeweled), aiming to blend fun with cognitive exercises. Especially designed for ease of use, they cater to older individuals, including those with dementia, gradually increasing in difficulty to match player skill levels. The GGG stands out by integrating game design with everyday cognitive tasks, offering a practical simulation of grocery shopping. Developed with older adult input, VibrantMinds aims to enhance cognitive health in seniors through engaging, meaningful gameplay, supporting its clinical trial's focus on cognitive wellness in the aging.
  Arms: VibrantMinds + Standard Care

SUMMARY:
Computer games are increasingly utilized as tools for studying cognitive skills, aging, individual differences, and development. They offer a unique advantage by presenting challenges that more closely mirror the complexities and demands of everyday tasks compared to traditional laboratory experiments, clinical tests, and standardized assessments. Our team took an innovative step in this direction by developing a suite of tablet-based games, titled VibrantMinds. These games, varying in type, are designed to measure diverse cognitive indicators, acting as proxies for assessments typically conducted using paper-and-pencil tests in clinical settings.

VibrantMinds games have been specifically crafted to be user-friendly and engaging for older adults, including those with dementia. Our studies have shown that these individuals not only find the games accessible but also exhibit measurable improvement in gameplay, suggesting potential benefits for cognitive skill training.

Building on this foundation, we are now poised to conduct an in-depth investigation into the actual effectiveness of serious computer games (SCGs) for cognitive enhancement and their application in real-world settings for older adults. This next phase of research will leverage the VibrantMinds platform to carry out studies aimed at validating software-defined indicators of cognitive function and measuring the impact of game-based interventions on cognitive abilities, health-related quality of life, and other significant real-life outcomes.

The anticipated results promise to expand our understanding of the potential for new technologies in cognitive assessment and intervention. Moreover, by employing machine learning analysis of the data collected through VibrantMinds, we aim to develop a taxonomy that correlates game complexity and player performance with conventional clinical instruments for assessing cognitive status and functioning.

ELIGIBILITY:
Inclusion Criteria:

* Older adults aged 65 years and older.
* Cognitive impairment within a specific range as measured by the Mini-Mental State -Examination (MMSE scores between 7 and 25).
* Ability to interact with the Serious Cognitive Games (SCGs) platform, indicating a necessary level of awareness.
* Functional vision and hearing, with or without aids (glasses/hearing aids), to engage with the SCGs platform.
* Functional upper extremity function to interact with the SCGs.

Exclusion Criteria:

* Presence of influenza, COVID-19, or another virus that could affect performance or pose a risk to others.
* Inability to communicate or comprehend instructions in English
* Moderate to severe limitations in upper extremity control or movement, significant visual or hearing impairments, or attention deficits that could impact the ability to successfully engage with the SCGs. Participants or their care partners who feel these conditions would interfere with study participation are excluded.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2022-08-03 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Cognition - Global | Baseline (Week 0), Post-Test (Week 12), Follow-up (Week 16)
  Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADASCog). Items are generally scored from 1-5; Final scores range 0-70, with higher scores indicating greater severity.

SECONDARY OUTCOMES:
Depression | Baseline (Week 0), Post-Test (Week 12), Follow-up (Week 16)
  Geriatric Depression Scale (GDS). Each Item is scored 0/1 (no/yes respectively), for a total of 15 questions, and a maximum of 15 points. Higher points indicate greater symptoms of depression.
Agitation | Baseline (Week 0), Post-Test (Week 12), Follow-up (Week 16)
  Cohen-Mansfield Agitation Inventory (CMAI). The CMAI is a 29 item scale, with each item ranging 1-7. Higher scores indicate greater agitation
Occupational Performance | Baseline (Week 0), Post-Test (Week 12), Follow-up (Week 16)
  The Canadian Occupational Performance Measure (COPM) employs a 1 to 10 scoring system, where clients rate their performance and satisfaction across chosen activities. A score of 1 indicates poor performance or satisfaction, while a score of 10 signifies excellent outcomes. Changes in these scores over time are used to evaluate the effectiveness of interventions based on client priorities.
Engagement | At each session from weeks 0-12; average 2x per week.
  Engagement questionnaire. A developed engagement questionnaire, with items ranked 1-5, will be utilized at each session
Affect | At each session from weeks 0-12; average 2x per week.
  The Positive and Negative Affect Schedule (PANAS) consists of two 10-item mood scales, measuring both positive and negative affect. Respondents rate each item on a scale from 1 (very slightly or not at all) to 5 (extremely), indicating the extent to which they have experienced each emotion. Higher scores represent greater positive or negative affect, respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- CapitalCare Group Inc Facilities, Edmonton, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: VibrantMinds Platform — https://vibrant-minds.org/vibrantminds2/start